CLINICAL TRIAL: NCT06208280
Title: An Exploratory Clinical Study to Evaluate the Safety and Tolerability of F01 in the Treatment of Autoimmune Diseases
Brief Title: F01 in the Treatment of Autoimmune Diseases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC 103-CD19CAR NK-103
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Diseases
Keywords: NK; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental)
  Interventions: Drug: After preconditioning with Fludarabine and Cyclophosphamide, F01 will be evaluated.

INTERVENTIONS:
Drug: After preconditioning with Fludarabine and Cyclophosphamide, F01 will be evaluated. — Drug: After preconditioning with Fludarabine and Cyclophosphamide, F01 will be evaluated.
  Biological: 0.5-3×10^9 CAR+NK Cells, Treatment follows a lymphodepletion Drug: Fludarabine: 25-30 mg/m^2 (D-5~D-3) Drug: Cyclophosphamide: 250-300 mg/ m^2 (D-5~D-3)

SUMMARY:
This is a multicenter, open lable clinical study to evaluate the safety and tolerability of F01 in autoimmune diseases.

DETAILED DESCRIPTION:
Approximately up to 20 participants with autoimmune diseases (including moderate-to-severe active systemic lupus erythematosus, relapse or refractory antineutrophil cytoplasmic antibody associated vasculitis,refractory idiopathic inflammatory myopathies and relapsed/refractory active diffuse cutaneous systemic sclerosis) are planned to enroll. This study is divided into two stages: dose escalation and dose extension.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be enrolled in the study:

Age ≥18 and ≤65 years old, gender unlimited.

Special criteria for different indications:

2.1 Patients with moderately to severely active SLE need to meet the following criteria：

Diagnosis of systemic lupus erythematosus (SLE) according to the European League Against Rheumatology/American College of Rheumatology (EULAR/ACR) SLE classification criteria (Aringer et al 2019) at least 6 months prior to screening.

Positive antinuclear antibody, and/or anti-double-stranded DNA antibody at screening.

Moderate to severe activity is defined as: SLEDAI 2000 score ≥ 8 points at screening Disease remains active after at least 2 months of use of standard SLE treatment regimen prior to screening.

Standard regimens for SLE include glucocorticoids and/or antimalarials, combined immunosuppressants/immunomodulators (including but not limited to azathioprine, mycophenolate mofetil, leflunomide, iratimod, methotrexate, cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, etc.), and/or biologic agents (including but not limited to rituximab, belimumab, telitacicept, etc.).

2.2 Patients with relapsed or refractory AAV should meet the following criteria：

Clinical diagnosis of granulomatosis with polyangitis (GPA) and microscopic polyangiitis (MPA) as defined by the 2012 Chapel Hill Consensus Conference (CHCC); At least one major item, or at least three other items, in Birmingham Vasculitis Activity Score (BVAS) version 3; Positive anti-protease-3 (PR3-ANCA) or antimyeloperoxidase (MPO-ANCA) at screening;

Relapsed/refractory is defined as:

Subjects with relapsed AAV: At least 1 disease recurrence (defined as the presence of at least one important item on the BVAS assessment, or at least 3 other items) after at least 3 months of treatment with glucocorticoids in combination with immunosuppressants (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.) (BVAS score 0 and glucocorticoid dose ≤ 7.5 mg/day prednisone or other equivalent glucocorticoid drugs) or 1-2 new items in two consecutive assessments), and disease recurrence occurred within 12 weeks prior to screening; Subjects with refractory AAV: Glucocorticoids combined with immunosuppressants (cyclophosphamide, rituximab, azathioprine, methotrexate, mycophenolate mofetil, etc.) for at least 3 months have not been effective (BVAS score of 0 and glucocorticoid dose ≤ 7.5 mg/day prednisone or other equivalent glucocorticoid drugs); 2.3 Patients with moderately to severely active IIM need to meet the following criteria： According to the 2017 EULAR/ACR classification criteria, the probability of diagnosing IIM is ≥55%, and it is classified as dermatomyositis (DM), polymyositis (PM), or immune-mediated necrotizing myopathy (IMNM) based on age at first onset, skin and muscle strength performance, laboratory tests, and muscle biopsy features;

Disease activity/severity meets the following criteria:

MMT-8 score ≤141 out of 150;

At least 2 of the other CSMs exceptions are met:

Patient-assessed overall activity (based on visual analogue scale (VAS) score≥2 points (range 0-10 points); Physician-assessed overall disease activity VAS score ≥2 points (range 0-10 points); Extramuscular global mobility VAS score ≥2 points (range 0-10 points); Health Assessment Questionnaire (HAQ) score ≥0.25 (range 0-3). At least 1 muscle enzyme level > 1.5 times ULN. - Prior intolerance or inadequate response to treatment with glucocorticoids and at least one other immunosuppressant or modulator, requiring that: Treatment with glucocorticoids and at least 2 immunosuppressants (azathioprine, methotrexate, mycophenolate mofetil, etc.) at known effective doses for at least 3 months; 2.4 Subjects with relapsed/refractory active diffuse cutaneous systemic sclerosis (dcSSc) need to meet the following criteria：

- Diagnosed systemic sclerosis according to the 2013 American College of Rheumatology/European Federation of Rheumatological Societies (ACR/EULAR) classification criteria for systemic sclerosis (SSc);

Consistent with diffuse cutaneous manifestations according to the criteria defined by LeRoy et al. 1988, i.e., extensive skin fibrosis with skin involvement of the elbow and/or proximal knee; Co-ordination of interstitial lung diseases (ILD) at screening with 45% predicted ≤ forced vital capacity (FVC) ≤ 70% predicted, or 40% predicted ≤ diffusing capacity of the lungs for carbon monoxide (DLCO) ≤ 70% predicted Relapsed/refractory is defined as relapse after failure to respond to conventional therapy or remission of disease.

Conventional treatment refers to the use of glucocorticoids, cyclophosphamide and at least one immunosuppressive/modulating drug for 6 months ≥, including azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, telitacicept, etc.

- Activity is defined as having at least one of the following: Evidence of skin progression at screening, i.e., a ≥10% increase in mRSS score in the last 6 months;

Evidence of activity in any of the following interstitial lung diseases (ILD) at screening:

Newly diagnosed ILD within the last 6 months; 10% reduction in FVC or 5% reduction in FVC with a 15% decrease in diffusing capacity of the lungs for carbon monoxide (DLCO) in participants with prior ILD in the last 6 months.

The expected survival is greater than 6 months.

Adequate bone marrow, liver, kidney, lung, cardiac, and coagulation function, defined as:

* Bone marrow function without blood transfusion and growth factor use within 7 days before routine blood: hemoglobin (Hb) ≥ 80 g/L, neutrophil count (ANC) ≥ 1.5×109/L, platelet count (PLT) ≥ 50×109/L;
* Renal function: creatinine clearance (CCr) ≥ 50 ml/min without hydration assistance, serum creatinine ≤ 1.5 times the upper limit of normal;
* Liver function: serum ALT and AST ≤ 2.5 times the upper limit of normal, total bilirubin ≤ 1.5 times the upper limit of normal;
* Lung function: Under indoor ventilation conditions, the blood oxygen saturation in the non-oxygen state is ≥ 92%; There was no clinically significant pleural effusion;
* Cardiac function: Left ventricular ejection fraction ≥ 40%; Echocardiography confirmed no clinically significant pericardial effusion., No clinically significant abnormalities were found in the ECG;

During the screening period, the serum pregnancy test results of fertile female subjects must be negative (women who have been surgically sterilized or have been menopausal for at least 2 years are considered not fertile). Fertile female subjects and male subjects must use highly effective contraceptive methods throughout the clinical study period and within 1 year after the last study treatment; At the same time, a commitment should be made not to donate eggs (egg cells, oocytes)/sperm for assisted reproduction within 1 year after the last study treatment.

Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will not be admitted to this clinical study:

Severe pulmonary disease in the past 1 year, such as moderate to severe pulmonary hypertension (echocardiographic mean pulmonary artery pressure > 60 mmHg), requiring oxygen storage mask oxygen therapy or non-invasive or invasive ventilator to assist breathing at screening Primary central nervous system lymphoma; SLE subjects need to exclude subjects who have had lupus crisis in the past 3 months, active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe neutropenia, severe myocardial damage, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, severe vasculitis;

Combined with severe kidney disease, including severe lupus nephritis, severe nephrotic syndrome, etc. Severe is defined as:

* Have received any of the following treatments within the specified time: Previous kidney transplantation; Dialysis or plasmapheresis within 3 months prior to screening; Pulse glucocorticoid therapy (defined as a dose ≥ 500 mg/d prednisone or equivalent dose of other glucocorticoids) within 1 month prior to screening;
* Need to receive either of the following treatments during the study: Need to use protocol prohibited medications; Need for dialysis or plasmapheresis; Kidney transplantation is required or planned.

History of severe cardiovascular disease, including but not limited to: symptomatic chronic heart failure requiring intervention, acute myocardial infarction in the past 6 months, unstable angina, history of severe arrhythmia, stroke; or New York Heart Association (NYHA) grade III~IV; History of other autoimmune diseases other than those for the target indication, including eosinophilic granulomatosis with polyangitis (EGPA), Henoch-Schoenlein purpura, rheumatoid arthritis, cryoglobulinemia vasculitis, inclusion body myositis (IBM), Anti-glomerular basement membrane disease, Behcet's disease or Takayasu's arteritis, etc; Family history of non-IIM myopathies such as drug-induced; myopathies, human immunodeficiency virus-associated myopathies, thyroid diseases, and myopathies; Patients with a history of malignancy, including tumor-related polymyositis/dermatomyositis. Patients who have been surgically resected and cured for non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, low-stage bladder cancer, ductal carcinoma in situ, or patients who have recovered without evidence of recurrence in the past two years and do not require treatment; Patients with known allergies, hypersensitivity, intolerance, or contraindications to F01 or any ingredient of drugs that may be used in the study (including fludarabine, cyclophosphamide, tocilizumab), or patients who have had a severe allergic reaction in the past;

Patients who have received the following treatments within the prescribed time frame prior tolymphodepletion pretreatment:

Received autologous/allogeneic hematopoietic stem cell transplantation or CAR-T and other cell therapy; Pulse glucocorticoid therapy within 2 months (defined as a dose of ≥500 mg/day prednisone or equivalent dose of other glucocorticoids); Have been treated with biologics such as belimumab or telitacicept within 1 month; Received major surgery, received live vaccine or received other clinical study treatment within 1 month; Presence of uncontrolled active infection requiring treatment with systemic antibiotics, antiviral, or antifungal drugs within 14 days, except for prophylactic therapy.

prednisone or equivalent glucocorticoids should be reduced to ≤20 mg/day at least 7 days before lymphodepletion Concomitant active hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus infection (HIV), or syphilis infection.

Risk of active tuberculosis at screening, regardless of completion of adequate treatment: presence of signs or symptoms of active tuberculosis (such as fever, cough, night sweats, and weight loss) as judged by the investigator at screening; Chest imaging (e.g., chest x-ray, chest CT scan) documented at screening or at any time within 6 months prior to screening showing active tuberculosis; Evidence of latent tuberculosis infection, such as a positive γ-interferon release test, at screening; Use of drug combinations/combination therapies prohibited by the protocol during screening; Any situations that the investigator believes the patients are not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with AEs and SAEs | Up to 12 weeks
  The incidence and severity of all adverse events, serious adverse events, and abnormal laboratory test results
The proportion of subjects with DLT | Up to 4 weeks
  Incidence of DLT

SECONDARY OUTCOMES:
Efficacy of F01 cells in autoimmune diseases | 24 weeks after infusion
  Proportion of SLE subjects with CR, LLDAS, and SRI-4 response(including SELENA-SLEDAI ≥4-Point improvement, BILAG 2004 with No new A domain score AND no more than 1 new B domain scores, PGA score increase less than 0.3 point from baseline)
Cellular kinetics | 96 weeks
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Ren Ji Hospital South Campus, School of Medicine, Shanghai JiaoTong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No